CLINICAL TRIAL: NCT07373613
Title: A Randomized, Multi-center, Double-Blind, Controlled, Parallel Design, Phase II Study to Evaluate the Efficacy and Safety Administration by Doses of BR1400-1, BR1400-2, BR1400-3, BR1400-4, and BR1400-5 in Patients With Essential Hypertension
Brief Title: A Study of BR1400-1, BR1400-2, BR1400-3, BR1400-4, and BR1400-5 in Patients With Essential Hypertension
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BR-FMS-CT-L202
Record Dates: First submitted 2026-01-20; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Essential Hypertension
MeSH Terms: conditions — Essential Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- BR1400-1 + BR1400-B + BR1400-C (Experimental): Patients will receive tablet BR1400-1 + BR1400-B (Placebo of BR1400-2 & BR1400-4)+ BR1400-C (Placebo of BR1400-5)
  Interventions: Drug: BR1400-1; Drug: BR1400-B; Drug: BR1400-C
- BR1400-A + BR1400-2 + BR1400-C (Experimental): Patients will receive BR1400-A (Placebo of BR1400-1 & BR1400-3) + BR1400-2 + BR1400-C (Placebo of BR1400-5)
  Interventions: Drug: BR1400-2; Drug: BR1400-A; Drug: BR1400-C
- BR1400-3 + BR1400-B + BR1400-C (Experimental): Patients will receive BR1400-3 + BR1400-B (Placebo of BR1400-2 & BR1400-4) + BR1400-C (Placebo of BR1400-5)
  Interventions: Drug: BR1400-3; Drug: BR1400-B; Drug: BR1400-C
- BR1400-A + BR1400-4 + BR1400-C (Experimental): Patients will receive BR1400-A (Placebo of BR1400-1 & BR1400-3) + BR1400-4 + BR1400-C (Placebo of BR1400-5)
  Interventions: Drug: BR1400-4; Drug: BR1400-A; Drug: BR1400-C
- BR1400-A + BR1400-B + BR1400-5 (Other): Patients will receive BR1400-A (Placebo of BR1400-1 & BR1400-3) + BR1400-B (Placebo of BR1400-2 & BR1400-4) + BR1400-5
  Interventions: Drug: BR1400-5; Drug: BR1400-A; Drug: BR1400-B
- BR1400-A + BR1400-B + BR1400-C (Placebo Comparator): Patients will receive BR1400-A (Placebo of BR1400-1 & BR1400-3) + BR1400-B (Placebo of BR1400-2 & BR1400-4) + BR1400-C (Placebo of BR1400-5)
  Interventions: Drug: BR1400-A; Drug: BR1400-B; Drug: BR1400-C

INTERVENTIONS:
Drug: BR1400-1 — One tablet administered alone
  Arms: BR1400-1 + BR1400-B + BR1400-C
Drug: BR1400-2 — One tablet administered alone
  Arms: BR1400-A + BR1400-2 + BR1400-C
Drug: BR1400-3 — One tablet administered alone
  Arms: BR1400-3 + BR1400-B + BR1400-C
Drug: BR1400-4 — One tablet administered alone
  Arms: BR1400-A + BR1400-4 + BR1400-C
Drug: BR1400-5 — One tablet administered alone
  Arms: BR1400-A + BR1400-B + BR1400-5
Drug: BR1400-A — One tablet administered alone
  Other Names: Placebo
  Arms: BR1400-A + BR1400-2 + BR1400-C; BR1400-A + BR1400-4 + BR1400-C; BR1400-A + BR1400-B + BR1400-5; BR1400-A + BR1400-B + BR1400-C
Drug: BR1400-B — One tablet administered alone
  Other Names: Placebo
  Arms: BR1400-1 + BR1400-B + BR1400-C; BR1400-3 + BR1400-B + BR1400-C; BR1400-A + BR1400-B + BR1400-5; BR1400-A + BR1400-B + BR1400-C
Drug: BR1400-C — One tablet administered alone
  Other Names: Placebo
  Arms: BR1400-1 + BR1400-B + BR1400-C; BR1400-3 + BR1400-B + BR1400-C; BR1400-A + BR1400-2 + BR1400-C; BR1400-A + BR1400-4 + BR1400-C; BR1400-A + BR1400-B + BR1400-C

SUMMARY:
The objective of this clinical trial is to evaluate the antihypertensive efficacy and safety of BR1400-1, BR1400-2, BR1400-3, BR1400-4, and BR1400-5 with essential hypertension.

ELIGIBILITY:
Inclusion Criteria:

<Screening Visit (V1)>

Patients with essential hypertension whose mean sitting systolic blood pressure (MSSBP) measured in the reference arm at the screening (Visit 1) meets the following criteria:

* For patients not currently receiving antihypertensive therapy: 140 mmHg ≤ MSSBP < 180 mmHg
* For patients receiving antihypertensive therapy : 130 mmHg ≤ MSSBP < 180 mmHg

For patients receiving antihypertensive therapy at the screening (Visit 1), those for whom the investigator determines that it is medically appropriate to temporarily discontinue their current antihypertensive treatment during the study.

<Baseline Visit (V2)>

Patients with essential hypertension whose mean sitting systolic blood pressure (MSSBP) measured in the reference arm at the baseline (Visit 2) prior to randomization meets the following criteria:

* For patients without cardiovascular disease: 140 mmHg ≤ MSSBP < 180 mmHg
* For patients with cardiovascular disease, diabetes with cardiovascular disease, albuminuria, or diabetes with chronic kidney disease (CKD): 130 mmHg ≤ MSSBP < 180 mmHg

Exclusion Criteria:

* Patients with blood pressure results showing MSSBP ≥ 180 mmHg or MSDBP ≥ 110 mmHg at screening(V1) and baseline(V2)
* Patients with a history of secondary hypertension or suspected secondary hypertension; (e.g., coarctation of the aorta, hyperaldosteronism, renal artery stenosis, renal hypertension, pheochromocytoma, Cushing's syndrome and polycystic kidney disease, etc.)
* Patients with shock
* Patients with orthostatic hypotension accompanied by symptoms

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to treatment of 8 weeks in MSSBP | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Hanyang University Hospital, Soeul, South Korea